CLINICAL TRIAL: NCT06664515
Title: Changes in Macular Pigment Optical Density After Full-thickness Macular Hole Closure Using Inverted Flap Technique
Brief Title: Changes InMPOD After Full-thickness Macular Hole Closure
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Ciro Costagliola, director, Federico II University
Other Study IDs: 05809853 Federico II
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Full Macular Hole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients affected by macular hole
  Interventions: Procedure: Ciro Costagliola

INTERVENTIONS:
Procedure: Ciro Costagliola — invert flap tecnique

SUMMARY:
The notable increase in MPOD following successful surgery suggests its potential role as a valuable adjunctive biomarker associated with a good visual prognosis following this type of macular hole surgical interventions.

DETAILED DESCRIPTION:
Full-thickness macular hole (FTMH) is a debilitating retinal disorder, particularly in its advanced forms, necessitating surgical intervention for vision restoration. This study showes the successful closure of a large FTMH using the inverted flap technique, highlighting the essential role of multimodal imaging, and particularly of macular pigment optical density (MPOD) assessment, in preoperative and postoperative evaluation.

Surgery was performed by an expert vitreoretinal surgeon, resulting in significant postoperative improvements in visual acuity and retinal architecture. Multimodal imaging, including MPOD assessment, played a pivotal role in preoperative evaluation and postoperative monitoring.

ELIGIBILITY:
Inclusion Criteria:age older than 60 years

* diagnosis of FTHM
* absence of other ocular diseases, responsible for macular edema (retinal vein occlusion, diabetic retinopathy, age-related macular degeneration

Exclusion Criteria:

No diagnosis of pseudophakic cystoid macular oedema

* previous treatment for pseudophakic cystoid macular oedema
* presence of other ocular diseases, responsible for macular edema (retinal vein occlusion, diabetic retinopathy, age-related macular degeneration)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The participans were older than 50 years with diagnosis of FTHM and underwent invert flap surgery.The participans did not present other ophthalmological diseases.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
MPOD After Full-thickness Macular Hole Closure (FTMH) | 6 months
  The parameters analyzed by OCT and MPOD six months after surgery are:
  OCT MPOD visual acuity
MPOD and Macula hole: before and after surgery | six months
  The parameters analyzed six months after surgery are:
  MPOD Visual acuity OCT

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Costagliola, Study Chair — FEDERICOII UNIVERSITY
Locations (1):
- University of Naples "Federico II", Naples, Italy, Italy